CLINICAL TRIAL: NCT00012103
Title: Prevention and Early Detection of Lung Cancer in Women
Brief Title: Computed Tomography for Early Detection of Cancer in Women Who Are at Risk for Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000068484; P30CA016087 (NIH); NYU-9928; NCI-G01-1913
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — Bronchoalveolar Lavage; Bronchoscopy

INTERVENTIONS:
Other: bronchoalveolar lavage
Other: screening questionnaire administration
Other: sputum cytology
Procedure: bronchoscopic and lung imaging studies
Procedure: bronchoscopy
Procedure: computed tomography
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Imaging procedures such as computed tomography may improve the ability to detect lung cancer earlier.

PURPOSE: Screening and diagnostic study of computed tomography in women who are at risk for lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability of computed tomography (CT) to detect early lung parenchymal abnormalities in women at high risk for lung cancer.
* Determine the number of abnormal findings detected by CT that develop into lung cancer in these patients.
* Correlate these abnormalities with the presence of K-ras and p53 mutations in the sputum and bronchoalveolar lavage in these patients.
* Develop and implement appropriate educational materials regarding lung cancer in women and provide referrals to other programs, such as smoking cessation programs.

OUTLINE: Patients complete a questionnaire at baseline to assess demographics, medical history, smoking history, menopausal status, estrogen therapy, and diet.

Patients then undergo a low-dose computed tomography (CT) scan without contrast. Patients with normal CT results undergo additional CT scans every 12 months.

Patients with abnormal CT results undergo a diagnostic CT scan (in the absence of prior studies). Patients with indeterminate nodules (less than 5 mm in size) undergo surveillance CT studies within 3-4 months. If nodules remain unchanged in size, patients undergo additional surveillance CT studies at 6 months and 1 year. Patients with lung parenchymal abnormalities on CT suspicious for malignancy undergo a bronchoscopy with biopsy and bronchoalveolar lavage (BAL). Patients with abnormal CT scan(s) and negative BAL for p53 and/or K-ras mutations or normal histology and positive BAL for K-ras and/or p53 mutations undergo additional CT scans at 6 months and 1 year. Patients with biopsy-proven malignancy after bronchoscopy are referred for definitive treatment.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Women who currently smoke or have smoking history of at least a 30 pack year

  * Pack year is defined by the number of pack(s) of cigarettes per day times the number of years of smoking
* No history of prior lung cancer

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior cancer within the past 5 years except basal cell or superficial skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Chachoua, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States